CLINICAL TRIAL: NCT01729572
Title: The Effect of add-on Tele Medicine Monitoring of Medication Adherence, on the Risk of Re-hospitalisation of Ambulatory Schizophrenic Patients. an Open, Prospective, Randomised Controled Trial
Brief Title: Measuring the Effect of Remote Monitoring of Treatment Adherence on the Risk of Re-admission of Ambulatory Schizophrenic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: SHL Telemedicine Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0004-12-SHA
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; Schizoaffective Disorder; disease management; treatment; rehabilitation; pharmacotherapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Tele-medicine monitoring (Experimental): Tele-medicine monitoring of medication adherence will be given to the study group as an add-on to routine out-patient treatment
  Interventions: Other: Tele-medicine monitoring of medication adherence
- No Intervention: Control Rutine out-patient treatment (No Intervention): routine out-patient treatment will be given to the control group

INTERVENTIONS:
Other: Tele-medicine monitoring of medication adherence
  Arms: Experimental: Tele-medicine monitoring

SUMMARY:
Schizophrenia is a chronic debilitating mental disorder, characterised by a relapsing remitting course. Although anti-psychotics can prevent relapse, its effect on schizophrenia outcome remains very limited, mainly due to very poor adherence to medications by the patients. This study aims to find, whether the add-on of remote monitoring of medication compliance via tele-medicine, to routine out-patient clinic care, can improve patients adherence and reduce the risk of relapse.

DETAILED DESCRIPTION:
Schizophrenia is a chronic debilitating mental disorder, characterised by a relapsing remitting course. Although anti-psychotics can prevent relapse, its effect on schizophrenia outcome remains very limited, mainly due to very poor adherence to medications by the patients. This study aims to find, whether the add-on of remote monitoring of medication compliance via tele-medicine, to routine out-patient clinic care, can improve patients adherence and reduce the risk of relapse. The study is an uni center, open, prospective, randomised and controlled.

ELIGIBILITY:
Inclusion Criteria:

* DSM 4 diagnosis of schizophrenia or schizoaffective
* able to give written informed consent
* Have a telephone line

Exclusion Criteria:

* Are not discharged to a place with routine medication monitoring
* Are not discharged under forced ambulatory treatment order
* Are not homeless
* Are not admitted due to drug intoxication or withdrawal.
* Are not admitted due to severe self harm.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Time to re-hospitalisation | 1 year
  Time to re-hospitalisation will be compared in the study group and in the control group during the follow-up period of up to one year

SECONDARY OUTCOMES:
number of re-hospitalisations | 1 year
  number of re-hospitalisations will be compared among the study and the control groups during the 1 year follow-up.

OTHER OUTCOMES:
Total time in hospital | 1 year
  Total time in hospital during the 1 year follow-up period will be compared between the study and the control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel